CLINICAL TRIAL: NCT07118956
Title: Respiratory-gated Transcutaneous Auricular Vagus Nerve Stimulation for Improving Apathy in Parkinson's Disease: A Randomized, Double-blind, Sham-controlled Trial
Brief Title: Respiratory-gated Transcutaneous Auricular Vagus Nerve Stimulation for Improving Apathy in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Head of the Department, Department of Neurology, The First Affiliated Hospital of Anhui Medical University, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PD-TaVNS-RCT
Record Dates: First submitted 2025-05-19; First posted 2025-08-12 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease; Apathy; Non-motor Symptoms; Vagus Nerve Stimulation
Keywords: Parkinson Disease; Apathy; Non-motor symptoms; Transcutaneous Auricular Vagus Nerve Stimulation
MeSH Terms: conditions — Parkinson Disease; Lethargy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active respiratory-gated transcutaneous auricular vagus nerve stimulation (RAVANS) (Experimental): Participants will receive active RAVANS daily for 2 week.
  Interventions: Other: Active RAVANS
- Sham RAVANS (Sham Comparator): Participants will receive sham RAVANS daily for 2 week.
  Interventions: Other: Sham RAVANS

INTERVENTIONS:
Other: Active RAVANS — Real RAVANS was performed on the cymba conchae of left ear in the vicinity of the auricular branch vagus nerve according to the Participant's respiratory rhythm. Stimulation parameters: frequency = 100 Hz; pulse width = 200 us, once a day, 30 minutes each time, one second of stimulation occurs during exhalation.
  Other Names: RAVANS
  Arms: Active respiratory-gated transcutaneous auricular vagus nerve stimulation (RAVANS)
Other: Sham RAVANS — Sham RAVANS was performed on on the cymba conchae of left ear according to the Participant's respiratory rhythm. Stimulation parameters: frequency = 100 Hz; pulse width = 200 us, once a day, 30 minutes each time, one second of stimulation occurs during exhalation and the interval between stimulus is 29 seconds.
  Other Names: RAVANS
  Arms: Sham RAVANS

SUMMARY:
The goal of this clinical trial is to learn whether 100HZ respiratory-gated vagus nerve stimulation (RAVANS) can improve the non-motor symptoms in people with Parkinson's disease (PD). It will also learn the safety of 100HZ RAVANS. The main questions it aims to answer are:

Can 100HZ RAVANS improve apathy in people with PD? Did the participants have any side effects or safety issues when undergoing 100HZ RAVANS? Researchers compared 100HZ RAVANS with sham stimulation (low-dose stimulation of the same site and treatment parameters) to see if 100HZ RAVANS could improve non-motor symptoms in patients with PD.

Participants will:

Receive 100HZ RAVANS or sham stimulation for 2 weeks. Neuropsychological assessment, imaging and biological sample collection were conducted before and after the entire cycle.

DETAILED DESCRIPTION:
This study employs a double-blind, sham-controlled design to further validate the effects of 100Hz RAVANS on apathy . Patients were randomized into real or sham stimulation groups. Both groups will receive RAVANS once daily, with each session lasting 30 minutes, for a total duration of two weeks. The study design will include neuropsychological assessments, imaging, and biological specimen collection before and after the entire cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for idiopathic Parkinson's disease (based on the MDS Clinical Diagnostic Criteria for Parkinson's Disease (2015 version)).
2. Patients with Apathy Motivation Index (AMI) score >1.7.
3. All PD patients must be on stable, standardized medication regimens with no adjustments to medications for at least 1 month prior to the study and throughout the study period.
4. Demonstrate good compliance and adherence, capable of completing behavioral tests and taVNS therapy.
5. Mini-Mental State Examination (MMSE) score ≥22.
6. Meet safety criteria for MRI screening.

Exclusion Criteria:

1. Prior brain MRI/CT showing focal brain lesions or severe white matter disease (Fazekas grade 3 or higher).
2. Secondary parkinsonism (e.g., vascular parkinsonism, drug-induced parkinsonism).
3. History of severe traumatic brain injury, neurosurgery, or deep brain stimulation (DBS) therapy.
4. Personal history of epilepsy, unexplained loss of consciousness, or current use of anticonvulsant medications for seizure control.
5. Diagnosis of neuropsychiatric disorders other than Parkinson's disease.
6. Current use of non-steroidal anti-inflammatory drugs (NSAIDs) or Non-benzodiazepine GABA receptor agonist drug or anticholinergics or corticosteroids, or history of substance abuse or drug addiction.
7. Participation in any clinical trial within the past 3 months.
8. Severe systemic comorbidities (e.g., hepatic/renal failure, arrhythmias, organic heart disease).
9. Pregnant/lactating women or subjects (including males) planning pregnancy within 6 months.
10. Contraindications to taVNS, such as cardiac pacemakers, post-DBS surgery, or auricular pathologies (e.g., tympanic membrane perforation).

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Apathy Motivation Index (AMI) | baseline; 2 weeks; 6weeks; 8weeks; 10 weeks
  The AMI is used to assess levels of apathy across behavioral, emotional, and cognitive domains. It provides a comprehensive measure of motivation deficits.

SECONDARY OUTCOMES:
Non-Motor Symptoms Scale, Second Version (NMSS-2) | baseline; 2 weeks; 6weeks; 8weeks; 10 weeks
  The NMSS-2 is a comprehensive, clinician-administered tool designed to assess the range and severity of non-motor symptoms in individuals with Parkinson's disease. It covers multiple domains including sleep disturbances, mood, cognition, gastrointestinal symptoms, urinary dysfunction, and other non-motor manifestations. This second version of the scale provides an updated and refined assessment framework to capture the broad impact of non-motor symptoms on patients' quality of life.
AMI subscales | baseline; 2 weeks; 6weeks; 8weeks; 10 weeks
  AMI has three subscale dimensions including behavioral activation, social motivation and emotional sensitivity.
Epworth Sleepiness Scale (ESS) | baseline; 2 weeks; 10 weeks
  The ESS is a widely used self-assessment questionnaire designed to measure daytime sleepiness. It was developed by Dr. Murray Johns in 1991 and is commonly employed in clinical and research settings to evaluate excessive daytime sleepiness , which is often associated with sleep disorders like obstructive sleep apnea ,narcolepsy, or insomnia.
Fatigue Scale-14 (FS-14) | baseline; 2 weeks; 10 weeks
  The FS-14 is a self-report measure used to evaluate fatigue across physical and mental dimensions. It comprises 14 items that assess the severity and impact of fatigue on daily functioning.
Pittsburgh Sleep Quality Index (PSQI) | baseline; 2 weeks; 10 weeks
  The PSQI is a standardized tool used to assess sleep quality and disturbances over a one-month time interval. It evaluates seven components of sleep, including subjective sleep quality, latency, duration, and daytime dysfunction.
REM Sleep Behavior Disorder Screening Questionnaire (RBDSQ) | baseline; 2 weeks; 10 weeks
  The RBDSQ is a diagnostic tool used to screen for REM Sleep Behavior Disorder (RBD), focusing on the presence of dream-enactment behaviors and other sleep-related symptoms.
The Unified Parkinson's Disease Rating Scale, Part III (UPDRS-III) | baseline; 2 weeks; 10 weeks
  The UPDRS-III is a standardized clinical assessment tool used to evaluate the motor symptoms of Parkinson's disease (PD). It is part of the broader UPDRS, which is the most widely accepted scale for assessing the severity and progression of PD. Below is a detailed explanation.
The Neuropsychiatric Inventory (NPI) | baseline; 2 weeks; 10 weeks
  The Neuropsychiatric Inventory (NPI) is a standardized tool used to assess neuropsychiatric symptoms (such as hallucinations, depression, agitation, etc.) in patients with dementia.
The Hamilton Anxiety Rating Scale (HAMA) | baseline; 2 weeks; 10 weeks
  The Hamilton Anxiety Rating Scale (HAMA) is a clinician-administered assessment tool widely used in clinical practice to evaluate the severity of anxiety symptoms
The Hamilton Depression Rating Scale (HAMD) | baseline; 2 weeks; 10 weeks
  The Hamilton Depression Rating Scale (HAMD) is a clinician-administered assessment tool commonly used in clinical practice to evaluate the severity of depressive symptoms.
Heart Rate Variability (HRV) | baseline everyday; during the intervention everyday
  Heart Rate Variability (HRV) is a physiological indicator that assesses the function of the autonomic nervous system (ANS) by analyzing subtle variations in heartbeat intervals (R-R intervals). The vagus nerve serves as the primary pathway of the parasympathetic nervous system. Transcutaneous auricular vagus nerve stimulation (taVNS) enhances parasympathetic nerve activity by stimulating the auricular branch of the vagus nerve. HRV is a critical metric for evaluating the efficacy of this regulatory effect.Each day before treatment, a 5-minute resting HRV is recorded, followed by a 30-minute HRV recording during the intervention.
Behavioral performance and computational parameters in an effort-based decision-making task | baseline; 2 weeks
  The Effort-Based Decision-Making Task is an experimental paradigm used to investigate how individuals weigh effort costs against task rewards under differenct conditions. Behavioral and computational indexes are calculated across varying levels of effort and reward.The main indicators are the selection rate and accuracy rate under different levels of effort and reward

CONTACTS AND LOCATIONS:
Overall Officials: Kai Wang, Ph.D., Principal Investigator — Anhui Medical University
Locations (1):
- Cognitive Neuropsychology Lab Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No